CLINICAL TRIAL: NCT05577949
Title: The Effect of Structured Aerobics Exercise Programme for the Improvement of Mental and Physical Health Parameters in Patients With Polycystic Ovary Syndrome: A Randomised Controlled Trial
Brief Title: Effect of Aerobics on Physical and Mental Health in Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Muhammad Irfan (Other)
Responsible Party: Sponsor-Investigator, Muhammad Irfan, Professor & Head, Department of Mental Health, Psychiatry and Behavioural Sciences, Peshawar Medical College
Organization: Peshawar Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aerobics & PCOs
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Structured aerobics exercise program; Physical health; Mental health
MeSH Terms: conditions — Polycystic Ovary Syndrome; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobics (Experimental): This group will perform structured aerobics exercise program in addition to the standard treatment given for women with PCOS.
  Interventions: Other: Structured aerobics exercise
- Management used as "Treatment As Usual" (No Intervention): This group will receive the standard management given for women with PCOS

INTERVENTIONS:
Other: Structured aerobics exercise — A 12 week structured aerobics exercise program will be offered. The patient has to perform exercise five times a week , 30 minutes a day
  Arms: Aerobics

SUMMARY:
Polycystic ovary is one of the most common metabolic and endocrine disorders in women of reproductive age group. The Rotterdam criteria are used internationally for its diagnosis. It has been reported that 57% of these women have at least one mental disorder. There is no health without mental health and it is fundamental to the good health and well-being of an individual. Women with PCOS are at risk of a wide range of significant psychological difficulties including depression, anxiety, eating disorders, sexual disorders, low self-esteem, poor body image, and overall low quality of life. In the healthy population, exercise plays a pivotal role in the optimization of mental health, but there is little evidence available to demonstrate its effects on women with PCOS. So, this study has been designed to study the effects of structured aerobics exercise programs on the mental and physical health of women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome is also referred to as "Hyperandrogenic anovulation or Stein Levinthal Syndrome". It has affected approximately 10 % of women of childbearing age. The prevalence of PCOS is higher among Pakistani women i.e. 52% as compared to the UK. The Rotterdam criteria are internationally used for the diagnosis of PCOS, which requires two out of the three features: signs of hyperandrogenism, ovulatory dysfunction, and ultrasound features of PCOS.

Although physical symptoms are increasingly recognized in women with PCOS, little attention has been paid to the mental health and well-being of these patients. PCOS creates an important psychological burden throughout the lifetime of these women. 57% of women with polycystic ovary syndrome have at least one mental disorder. Also, mental health is an essential part of public health and it is one of the most important indicators of the quality of health care in society.

Women with PCOS are at risk of a wide range of significant psychological difficulties including depression, anxiety, eating disorders, sexual disorders, low self-esteem, poor body image, and overall a lowered quality of life. In a healthy population, lifestyle modifications, particularly physical activity, and exercise play a pivotal role in the optimization of mental health but there is little evidence available to demonstrate the effects of exercise on the optimization of psychological well-being and physical health of women with PCOS. So, this study has been designed to study the effect of a structured aerobics exercise program on the mental and physical health of women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

All women diagnosed with PCOS according to the Rotterdam criteria with the age range of 18-49 years

Exclusion Criteria:

1. Women that do not own personal smartphones
2. Patients with endocrinological diseases like diabetes mellitus
3. Thyroid, adrenal, or pituitary dysfunction
4. Hepatic and pulmonary diseases
5. Orthopedic
6. Other diseases which can limit their physical activity or make it hazardous for them
7. Participants with significant cognitive impairment, like intellectual disability or dementia, or active psychosis.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
PCOS Quality of Life scale | 12 weeks (3 months)
  Change in the score of the PCO quality of life scale from baseline to midway to end of therapy, higher scores mean a better quality of life.
Hospital Anxiety and Depression Scale | 12 weeks (3 months)
  Change in the score of the Hospital anxiety and depression scale from baseline to midway to end of therapy, 0-7 indicates normal, 8 to 10 indicates borderline and 11-21 indicates abnormal cases. Higher scores mean a worse outcome

SECONDARY OUTCOMES:
ENRICH marital satisfaction scale | 12 weeks (3 months)
  Change in the score of the ENRICH marital satisfaction scale from baseline to midway to end of therapy, higher scores mean better marital satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Kareem, MBBS,FCPS, Principal Investigator — Peshawar Medical College
Locations (4):
- Pakistan (4):
  - Hayatabad Medical Complex, Peshawar, Khyber Pakhtunkhwa
  - Khyber teaching hospital, Peshawar, Khyber Pakhtunkhwa
  - Northwest teaching hospital and research centre, Peshawar, Khyber Pakhtunkhwa
  - Mercy teaching hospital, Peshawar, Khyber Pukhtunkhwa

IPD SHARING:
Plan to Share IPD: No